CLINICAL TRIAL: NCT00842504
Title: Alternate Day Micafungin Anti-Fungal Prophylaxis in Immunocompromised Pediatric Patients: A Pharmacokinetic Study
Brief Title: Alternate Day Micafungin: A PK Study in Pediatric Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Micafungin PK
Record Dates: First submitted 2009-02-11; First posted 2009-02-12 (Estimated); Last update posted 2012-02-16 (Estimated); Status verified 2012-02

CONDITIONS: Fungal Infection
Keywords: Anti-fungal; Immunocompromised; Pharmacokinetic; Prophylaxis; Pharmacokinetics
MeSH Terms: conditions — Mycoses | interventions — Micafungin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Micafungin (Other): 3 mg/kg given once
  Interventions: Drug: Micafungin

INTERVENTIONS:
Drug: Micafungin — 3 mg/kg IV once over 1 hour
  Other Names: MYCAMINE

SUMMARY:
The purpose of this study is to examine the pharmacokinetics of micafungin when it is given on an every other day schedule. The study will determine if every other day micafungin will provide drug exposure equivalent to daily dosing while reducing administration costs and improving patient convenience. Fifteen patients will be enrolled on this study. Blood samples for PK measurements will be obtained for 48 hours following a single dose of micafungin (3 mg/kg).

DETAILED DESCRIPTION:
Disseminated fungal infection is a major cause of morbidity and mortality in immunocompromised children. Many of the drugs used for fungal prophylaxis have been associated with kidney and liver toxicity. Also, breakthrough infections have been reported with the use of some of the oral agents due to poor oral absorption. An alternative approach is the use of intravenous micafungin for fungal prophylaxis. Micafungin has a distinct advantage due to its better safety profile, specifically in terms of liver and kidney toxicity. Currently, children who receive micafungin are given daily dosing. This study will examine the pharmacokinetics of micafungin when it is given on an every other day schedule. It will examine whether every other day micafungin will provide drug exposure equivalent to daily dosing while reducing administration costs and improving patient convenience. Both animal and adult human data support the use of this approach. Fifteen patients will be enrolled on this study and will be given a single dose of micafungin (3 mg/kg). Blood samples will be drawn for pharmacokinetic measurements after administration of micafungin.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized patients who are at risk for fungal infection and require prophylaxis.
* Age ≤ 10 years excluding neonates
* Children must have an indwelling venous access device
* Patients with adequate organ function (documented within 2 weeks prior to start of micafungin): creatinine < 2 times upper limit normal; ALT, AST and total bilirubin ≤ 3 times upper limit normal

Exclusion Criteria:

* Patients who are < 28 days old (neonates) or > 10 years of age
* Patients who have history of past or evidence of active fungal disease (by either radiological studies or biopsy proven) or are being treated for presumed fungal infection.
* Patients who have history of allergy to micafungin or other echinocandin preparations, such as Caspofungin or Anidulafungin.
* Patients who have received micafungin or other echinocandin preparations in the previous two weeks.
* Patients receiving antifungal prophylaxis other than Fluconazole at the time of enrollment.
* Failure to sign informed consent, or inability to undergo informed consent process.
* Not medically advisable to obtain the specimens necessary.

Ages: 29 Days to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15 (Actual)
Dates: Start 2007-07; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Every other day micafungin will provide drug exposure equivalent to daily dosing while reducing administration costs and improving patient convenience. | 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Parinda Mehta, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States